CLINICAL TRIAL: NCT05923879
Title: Mechanism Investigation of Selinexor Combined With Lenalidomide and Rituximab in the Treatment of Diffuse Large B-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Other Study IDs: SR2-DLBCL
Record Dates: First submitted 2023-06-03; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Selinexor combined with lenalidomide and rituximab — Selinexor combined with lenalidomide and rituximab

SUMMARY:
This is a retrospective observational study of the therapeutic mechanism and resistance mechanism of the treatment of Selinexor combined with lenalidomide and rituximab in diffuse large B-cell lymphoma patients. By detecting the immune cells in peripheral blood and tumor tissues of patients before and after treatment, the key immune cell subsets and immune molecules linked to the action and resistance of the treatment of Selinexor combined with lenalidomide and rituximab, so as to provide the basis for the optimization of the treatment or the combination of other immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Histopathologically confirmed diffuse large B-cell lymphoma according to World Health Organization (WHO) classification criteria 2016.
3. There is evidence of relapsed or refractory disease.
4. Treatment with Selinexor combined with lenalidomide and rituximab.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18-year-old recurrent or refractory diffuse large B-cell lymphoma patients receiving Selinexor combined with lenalidomide and rituximab would be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor tissues collected before treatment and at the point of progression if available for DNA sequencing after quality control. | 2023/06/30-2025/06/30
  Tumor tissues collected before treatment and at the point of progression if available for DNA sequencing after quality control. On the one hand, the difference of tumor mutations will be analyzed in pre-treatment biopsy samples of patients grouped by efficacy; on the other hand, the changes of tumor mutations will be analyzed between pre-treatment and post-treatment biopsy samples of patients.
Tumor tissues collected before treatment and at the point of progression if available for RNA sequencing after quality control. | 2023/06/30-2025/06/30
  Tumor tissues collected before treatment and at the point of progression if available for bulky RNA sequencing, single-cell RNA sequencing and spatial transcriptome sequencing after quality control. On the one hand, the difference of characteristics of tumor microenvironment will be analyzed in pre-treatment biopsy samples of patients grouped by efficacy; on the other hand, the changes of characteristics of tumor microenvironment will be analyzed between pre-treatment and post-treatment biopsy samples of patients.
Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023/06/30-2025/06/30
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and chemokines and cytokines.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided